CLINICAL TRIAL: NCT04784377
Title: High Intensity Versus Low Level Laser Therapy in Treatment of Patients With Subacromial Impingement Syndrome: A Randomized, Double-blind, Controlled Trial.
Brief Title: High and Low Laser for Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser and impingement syndrome
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2021-03

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High laser group (Experimental)
  Interventions: Other: high intensity laser in addition to traditional physical therapy exercises
- low laser group (Experimental)
  Interventions: Other: low level laser in addition to traditional physical therapy exercises
- control group (Other)
  Interventions: Other: traditional physical therapy exercises

INTERVENTIONS:
Other: high intensity laser in addition to traditional physical therapy exercises — high intensity laser will be used with 1064 nm wavelength and maximum of 25 W power. Analgesic and biostimulant modes were used in the present study.
  Also the patients will receive traditional physical therapy exercises in the form of flexibility and strengthening exercises for shoulder muscles.
  Arms: High laser group
Other: low level laser in addition to traditional physical therapy exercises — patients will receive low level Laser Therapy in addition to traditional physical therapy exercises.
  diode laser device with a wavelength of 850nm, power output of 100mV, continuous wave and 0.07cm2 spot area laser will be used. The laser will be applied with a dosage of 5 joule/cm2 (totally 15-20 joule) at the most 5 painful points for 1 minute at each point over subacromial region of the shoulder.
  Also the patients will receive traditional physical therapy exercises in the form of flexibility and strengthening exercises for shoulder muscles.
  Arms: low laser group
Other: traditional physical therapy exercises — Also the patients will receive traditional physical therapy exercises in the form of flexibility and strengthening exercises for shoulder muscles.
  Arms: control group

SUMMARY:
Shoulder pain is the third most common musculoskeletal problem after lumbar and neck diseases in clinical practice, and the most common cause of shoulder pain is subacromial impingement syndrome. The main goal of treatment is to reduce pain and to solve the mechanical problem that causes functional impairment. Low-level laser treatment is an increasingly used treatment modality in the treatment of subacromial impingement syndrome as in many musculoskeletal diseases, as it promotes cell proliferation and tissue regeneration by its anti-inflammatory and photobiostimulation properties. Also, High-intensity laser therapy is a treatment method that is gaining popularity in the recent years. These ultra-short impulses effect a deep action in the biological tissue (3-4 cm), with a homogeneous distribution of the light source in the irradiated soft tissue, but without excessive thermal enhancements. It reduces pain and edema with photomechanic effects in deep tissues. As far as the investigators know, there are no studies comparing these two treatment modalities in subacromial impingement syndrome yet. This study was planned to compare the efficacy of High-intensity laser therapy and low-intensity laser therapy in treatment of patients with subacromial impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain for at least one month
* male and female patients with age range from 25-45 years old
* positive impingement test results
* stage I or II disease according to the Neer classification, confirmed by MRI
* visual analog scale score greater than 40 mm.

Exclusion Criteria:

patients will be excluded if they have:

* major trauma to the shoulder
* stage III subacromial impingement syndrome
* diabetes mellitus
* hypothyroidism
* calcific tendinitis
* adhesive capsulitis (forward flexion less than 160, horizontal abduction less than 160
* installation of cardiac pacemaker
* history of a physical therapy program for the same shoulder in the last 6 months.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
pain intensity | change from base line at three weeks
  Pain will be evaluated by a visual analogue scale (VAS). The patient will be asked to mark the severity of pain on a 100-mm line with "no pain" on one end and "most unbearable pain" on the other end

SECONDARY OUTCOMES:
shoulder range of motion | change from baseline at three weeks
  Flexion, abduction, and external rotation will be measured by using goniometer in a supine position and the active movements will be recorded. The goniometer will be centered at the acromion for abduction, greater tubercle for flexion, and olecranon for external rotation at 90° shoulder and elbow flexion
pain pressure threshold | change from baseline at three weeks
  Pressure Pain Threshold will be determined with an analogue algometer at the most painful point of the subacromial area. This point will be determined by a previous examination based on the point that the patient determined as 'his or her point of maximum pain'.
Shoulder Pain and Disability Index | change from baseline at three weeks
  this scale will be used to assess functional status of the shoulder. The SPADI includes shoulder questions and consists of two subscales: pain and disability. Pain subscale consists of 5 items, and disability subscale consists of 8 items, and the total score is 0-100
Pittsburgh Sleep Quality Index (PSQI) | change from baseline at three weeks
  This scale assesses sleep quality and disorder and consists of seven subcomponents (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, drug use, and daytime functions) and 19 items. Each component is evaluated on a score of 0-3 and is evaluated with a total sleep score ranging from 0 to 21, and high scores represent low sleep quality. A PSQI total score < 5 points is considered "good" sleep quality and > 5 points is "bad" sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

REFERENCES:
- [Background] Bal A, Eksioglu E, Gurcay E, Gulec B, Karaahmet O, Cakci A. Low-level laser therapy in subacromial impingement syndrome. Photomed Laser Surg. 2009 Feb;27(1):31-6. doi: 10.1089/pho.2007.2222. PMID 19250050
- [Background] Alfredo PP, Bjordal JM, Junior WS, Marques AP, Casarotto RA. Efficacy of low-level laser therapy combined with exercise for subacromial impingement syndrome: A randomised controlled trial. Clin Rehabil. 2021 Jun;35(6):851-860. doi: 10.1177/0269215520980984. Epub 2020 Dec 14. PMID 33307783
- [Background] Aceituno-Gomez J, Avendano-Coy J, Gomez-Soriano J, Garcia-Madero VM, Avila-Martin G, Serrano-Munoz D, Gonzalez-Gonzalez J, Criado-Alvarez JJ. Efficacy of high-intensity laser therapy in subacromial impingement syndrome: a three-month follow-up controlled clinical trial. Clin Rehabil. 2019 May;33(5):894-903. doi: 10.1177/0269215518824691. Epub 2019 Jan 23. PMID 30672303